CLINICAL TRIAL: NCT04503850
Title: Impact of Beta 3 Agonist Mirabegron on Erectile Function on Patients With Benign Prostate Hyperplasia
Brief Title: Impact of Mirabegron on Erectile Function in BPH Patients
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Kasr El Aini Hospital (Other)
Responsible Party: Principal Investigator, Samer Morsy, Urology Consultant, Kasr El Aini Hospital
Other Study IDs: Cairo University Hospitals
Record Dates: First submitted 2020-08-03; First posted 2020-08-07 (Actual); Last update posted 2020-08-10 (Actual); Status verified 2020-08

CONDITIONS: Males With Benign Prostatic Hyperplasia Symptoms
MeSH Terms: interventions — mirabegron; Adrenergic alpha-Antagonists

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Group A Mirabegron: 50 patients receiving Mirabegron 50 mg once daily & alpha blocker
  Interventions: Drug: Mirabegron 50 MG
- Group B alpha blocker only: 50 patients receiving alpha blocker only
  Interventions: Drug: Alpha Blockers

INTERVENTIONS:
Drug: Mirabegron 50 MG — Mirabegron 50 mg daily dose and follow Up of erectile function using international index of erectile function 5 scoring system
  Groups: Group A Mirabegron
Drug: Alpha Blockers — Alpha blocker daily and evaluation of erectile function using international index of erectile function 5 scoring system
  Groups: Group B alpha blocker only

SUMMARY:
Evaluation of impact of Mirabegron on erectile function for patients treated for BPH

DETAILED DESCRIPTION:
50 patients (Group A) will receive Mirabegron & alpha blocker 50 patients (Group B) will receive alpha blocker only Evaluation using IIEF 5 scoring system

ELIGIBILITY:
Inclusion Criteria:

* All males above age 50 with LUTS due to BPH not candidate for prostatectomy

Exclusion Criteria:

* males below age 50
* neurologic abnormality
* Any indication for prostatectomy
* abnormal bladder contractility i.e diabetics

Min Age: 50 Years | Sex: Male
Age Groups: Adult, Older Adult
Study Population: All males above age of 50 with LUTS due to BPH
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2020-10-01 (Estimated); Primary Completion 2021-05-01 (Estimated); Study Completion 2021-10-01 (Estimated)

PRIMARY OUTCOMES:
Impact of Mirabegron on erectile function | 6 months
  Using international index of erectile function 5 score system , least score 5 means severe erectile dysfunction and highest score 25 means no erectile dysfunction

IPD SHARING:
Plan to Share IPD: Undecided